CLINICAL TRIAL: NCT07300150
Title: A Phase 1, Open-label Dose Escalation and Expansion Study OF PT0511 in Participants With KRAS Mutated OR Amplified Advanced Solid Tumors
Brief Title: A Study of PT0511 in Participants With KRAS Mutated or Amplified Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: PAQ Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PT0511-101
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer; Pancreatic Cancer; Non-Small Cell Lung Cancer; Solid Tumor
Keywords: KRAS
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (9):
- Part 1a: Dose Escalation (Experimental): Participants with solid tumors with any KRAS mutation or amplified WT KRAS will receive PT0511 infusion, intravenously (IV), until disease progression or intolerance.
  Interventions: Drug: PT0511
- Part 1b: Dose Expansion: Tumor type 1 (Experimental): Participants with tumor type 1 will receive PT0511 infusion until disease progression or intolerance. Recommended dose or doses for expansion for Part 1b will be determined based on the safety, tolerability, pharmacokinetic (PK) and pharmacodynamic (PD) data for PT0511 established in Part 1a.
  Interventions: Drug: PT0511
- Part 1b: Dose Expansion: Tumor type 2 (Experimental): Participants with tumor type 2 will receive PT0511 infusion in combination with cetuximab infusion, until disease progression or intolerance. Recommended dose or doses for expansion for Part 1b will be determined based on the safety, tolerability, PK and PD data for PT0511 established in Part 1a.
  Interventions: Drug: PT0511; Drug: Cetuximab
- Part 1b: Dose Expansion: Tumor type 3 (Experimental): Participants with tumor type 3 will receive PT0511 infusion until disease progression or intolerance. Recommended dose or doses for expansion for Part 1b will be determined based on the safety, tolerability, PK and PD data for PT0511 established in Part 1a.
  Interventions: Drug: PT0511
- Part 1b: Dose Expansion: Tumor type 4 (Experimental): Participants with tumor type 4 will receive PT0511 infusion until disease progression or intolerance. Recommended dose or doses for expansion for Part 1b will be determined based on the safety, tolerability, PK and PD data for PT0511 established in Part 1a.
  Interventions: Drug: PT0511
- Part 1b: Dose Expansion: Tumor type 5 (Experimental): Participants with tumor type 5 will receive PT0511 infusion until disease progression or intolerance. Recommended dose or doses for expansion for Part 1b will be determined based on the safety, tolerability, PK and PD data for PT0511 established in Part 1a.
  Interventions: Drug: PT0511
- Part 1b: Dose Expansion: Tumor type 6 (Experimental): Participants with tumor type 6 will receive PT0511 infusion until disease progression or intolerance. Recommended dose or doses for expansion for Part 1b will be determined based on the safety, tolerability, PK and PD data for PT0511 established in Part 1a.
  Interventions: Drug: PT0511
- Part 1b: Dose Expansion: Tumor type 7 (Experimental): Participants with tumor type 7 will receive PT0511 infusion until disease progression or intolerance. Recommended dose or doses for expansion for Part 1b will be determined based on the safety, tolerability, PK and PD data for PT0511 established in Part 1a.
  Interventions: Drug: PT0511
- Part 1b: Dose Expansion: Tumor type 8 (Experimental): Participants with tumor type 8 will receive PT0511 infusion until disease progression or intolerance. Recommended dose or doses for expansion for Part 1b will be determined based on the safety, tolerability, PK and PD data for PT0511 established in Part 1a.
  Interventions: Drug: PT0511

INTERVENTIONS:
Drug: PT0511 — Intravenous infusion.
Drug: Cetuximab — Intravenous infusion.
  Arms: Part 1b: Dose Expansion: Tumor type 2

SUMMARY:
The primary purpose of this study is to evaluate the safety and tolerability, determine the maximally tolerated dose (MTD) and/or recommended Phase 2 dose(s) (RP2D) of PT0511 in adult participants with solid tumors as monotherapy and in combination with cetuximab in participants with colorectal cancer (CRC).

ELIGIBILITY:
Inclusion Criteria:

1. Men or women >=18 years of age
2. Histologically or cytologically confirmed advanced or metastatic solid malignancy.
3. Participant has a pathologically documented, locally advanced or metastatic malignancy with any KRAS mutation or wild-type (WT) KRAS amplification identified through molecular testing using a Clinical Laboratory Improvement Amendments (CLIA) certified, validated institutional or commercial test.

   • Participant must have received at least 1 and no more than 4 prior systemic therapies or be intolerant or ineligible for available therapies known to provide clinical benefit.
4. Measurable disease (RECIST 1.1 Criteria).
5. ECOG Performance Status 0 or 1.
6. Willingness to avoid pregnancy or fathering children screening through 90 days after the last dose of study treatment.

Exclusion Criteria:

Cancer History

1. Active brain metastasis or carcinomatous meningitis. If participants have had brain metastases resected or have received radiation therapy, they may be eligible if: (1) study treatment begins at least 4 weeks from the end of brain-specific therapy, (2) residual neurological symptoms Grade <=2, (3) currently on stable doses of corticosteroids, and (4) pre-study brain MRI documents no new/worsening brain lesions.
2. History of any other malignancy within the past 2 years, except:

   * Malignancy treated with curative intent and with no known active disease present >=2 years before enrolment and felt to be at low risk for recurrence by the investigator.
   * Basal or squamous cell carcinoma of the skin, in situ cervical cancer, early -stage endometrial cancer that has been definitively treated, superficial bladder cancer, Gleason 6/7 treated prostate cancer, and ductal carcinoma in situ or lobular carcinoma in situ of the breast.

   Prior Cancer Therapy
3. Unresolved toxicities from prior anti-cancer therapies. Participants with prior endocrine replacement therapies are eligible for entry even if administered to treat endocrine deficiency due to the prior anti-cancer therapy.
4. Concurrent participation in another interventional clinical study.
5. Treatment with anticancer medications or investigational drugs within the following intervals before the first administration of study drug:

   * At least 14 days for chemotherapy or targeted small-molecule therapy.
   * At least 28 days for a prior monoclonal antibody.
   * At least 28 days or 5 half-lives (whichever is longer) for all other investigational study drugs or devices. For drugs with very long half-lives, participants may be allowed to enroll prior to 5 half-lives at the discretion of the investigator in discussion with the medical monitor.
   * Note: Concurrent hormonal therapy for prostate or breast cancer is allowable
6. Prior treatment with a KRAS/RAS degrader.

   Medical History
7. Significant cardiovascular disease within 6 months of starting study therapy.
8. Active infection requiring antibiotics within 7 days of study treatment.
9. Known HIV infection with a CD4+ T-cell count <200 cells/mcL and/or a detectable viral load per parameters of assay and/or on an anti-retroviral regimen containing a strong or moderate CYP3A4/5 inhibitor or inducer and/or on a new anti-retroviral regimen for less than 28 days prior to the initiation of study treatment.
10. Known history of drug-induced liver injury; primary biliary cirrhosis; or ongoing extrahepatic obstruction caused by stones, cirrhosis of the liver, or portal hypertension.
11. Major surgery within 4 weeks of the start of study therapy or postoperative complications preventing the participant from adhering to protocol assessments and procedures.
12. Known hypersensitivity to any of the products to be administered during dosing.
13. Any disease or disorder that, in the opinion of the investigator, may compromise the ability of the participant to provide written informed consent and/or to comply with all required study procedures.

    Medications
14. Part 1a (Dose escalation): Use of a strong or moderate CYP3A4/5 inhibitor or inducer, Use of a strong P-gp inhibitor or inducer.

    Organ Function
15. Participants with laboratory values indicating inadequate hematology, hepatic, or renal function.

    Diagnostic Assessments
16. Clinically significant abnormalities in rhythm, conduction, or morphology of resting ECG.
17. Baseline QT interval corrected for heart rate using Fridericia's formula (QTcF) >=470 msec
18. Female participants of childbearing age with a positive urine or serum test within 7 days of study start or confirmation from Ob/Gyn that any positive bHCG test is not representative of an ongoing pregnancy.
19. Women who are lactating/breast feeding or who plan to breastfeed while on study through 28 days after receiving the last dose of study drug.
20. Active HBV infection. Participants with resolved infection or who are on Stable antiviral therapy are eligible.
21. Active HCV infection. Participants who have completed definitive antiviral therapy with post treatment confirmation of eradication are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2028-10-18 (Estimated); Study Completion 2028-10-18 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose-limiting Toxicities (DLT) | Cycle 1 (Cycle length=21 days)
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | Up to 24 months
Number of Participants with TEAEs Leading to Treatment Interruptions, Dose Reductions and Permanent Discontinuations | Up to 24 months

SECONDARY OUTCOMES:
Cmax/C0: Maximum Blood Concentration (Cmax) and/or Concentration at Time 0 (C0) of PT0511 | Cycle 1 Days 1 and 15: Pre-infusion and up to 24 hours post-infusion (Cycle length=21 days)
Tmax: Time to Reach Cmax of PT0511 | Cycle 1 Days 1 and 15: Pre-infusion and up to 24 hours post-infusion (Cycle length=21 days)
AUC0-t: Area Under the Curve From time 0 to the time of the Last Quantifiable Concentration of PT0511 | Cycle 1 Days 1 and 15: Pre-infusion and up to 24 hours post-infusion (Cycle length=21 days)
t1/2: Terminal Elimination Half-life of PT0511 | Cycle 1 Days 1 and 15: Pre-infusion and up to 24 hours post-infusion (Cycle length=21 days)
AUC0-∞: Area Under the Curve From Time 0 Extrapolated to Infinity of PT0511 | Cycle 1 Days 1 and 15: Pre-infusion and up to 24 hours post-infusion (Cycle length=21 days)
CL: Clearance of PT0511 | Cycle 1 Days 1 and 15: Pre-infusion and up to 24 hours post-infusion (Cycle length=21 days)
Vd: Volume of Distribution of PT0511 | Cycle 1 Days 1 and 15: Pre-infusion and up to 24 hours post-infusion (Cycle length=21 days)
Overall Response Rate (ORR) | Up to 12 months
  ORR will be determined by radiographic disease assessments per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Duration of Response (DOR) | Up to 12 months
  DOR will be determined by radiographic disease assessments per RECIST 1.1.
Number of Participants with Antitumor Activity Markers in Peripheral Blood of PT0511 | Cycle 1 Day 15: Pre-infusion and up to 24 hours post-infusion (Cycle length=21 days)
Overall Survival (OS) | At 1 year
  OS is defined as the time from enrollment up to death due to any cause.
Progression-free Survival (PFS) | At 1 year
  PFS will be determined by radiographic disease assessments per RECIST 1.1.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Dana-Farber/Massachusetts General Hospital, Inc, Boston, Massachusetts
  - New Experimental Therapeutics of San Antonio LLC, San Antonio, Texas
  - START - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
  - START Mountain Region, West Valley City, Utah
  - NEXT Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Yes